CLINICAL TRIAL: NCT06367634
Title: A Prospective, Multi-Center, Randomized, Controlled, Subject- and Evaluator-Blinded, Non-Inferior Clinical Investigation of the Safety and Effectiveness of TEOSYAL® PureSense ULTRA DEEP Versus Restylane® Lidocaine for the Correction of Moderate to Severe Nasolabial Folds in Chinese Adults
Brief Title: TEOSYAL® PureSense ULTRA DEEP Versus Restylane® Lidocaine for the Correction of Moderate to Severe Nasolabial Folds in Chinese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEO-TSUL-2301
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Nasolabial Folds
Keywords: Dermal Filler; Hyaluronic Acid
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded-Live evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra Deep (Experimental)
  Interventions: Device: injection in NLF
- Restylane (Active Comparator)
  Interventions: Device: injection in NLF

INTERVENTIONS:
Device: injection in NLF — TEOSYAL® PureSense ULTRA DEEP is a sterile, transparent, non-pyrogenic, viscoelastic gel made of HA of non-animal origin

SUMMARY:
This is a prospective, multi-center, randomized, controlled, subject- and evaluator-blinded clinical investigation to demonstrate non-inferiority of TEOSYAL® PureSense ULTRA DEEP compared to Restylane® Lidocaine for the correction of moderate to severe NLF in Chinese adults.

Eligible subjects will be enrolled and randomized either to the treatment group or control group in a 1:1 ratio on Day 0. Each subject assigned to the treatment group will receive TEOSYAL® PureSense ULTRA DEEP in both NLFs, whereas subjects assigned to the control group will receive Restylane® Lidocaine.

The treating investigator will administer the corresponding product in both NLFs of the subject on Day 0.

All subjects will return to the site at 4, 12, 24, 36, and 52 weeks after the last treatment for effectiveness and safety assessment. All subjects will receive a safety phone call 7 days after the initial treatment at baseline, and after the touch-up treatment, if applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male and female, 18 years of age or older.
2. Subject desiring bilateral NLF treatment.
3. Has symmetrical NLFs, with the same WSRS score of 3 (moderate) or 4 (severe) for both right and left NLFs, as determined on live assessment by the blinded evaluator.
4. Subject willing to abstain from all other facial aesthetic procedures/therapies that could interfere with effectiveness evaluations (e.g., dermal fillers outside of this investigation, toxin treatments, facial ablative or fractional laser, intense pulsed light [IPL], microdermabrasion, chemical peels, skin bleaching agents, non-ablative laser, or energy-based device for skin-tightening, surgical procedures, etc.) during participation in the investigation.
5. Woman of childbearing potential must be using a highly effective method of birth control .
6. Subject understands and is able to follow instructions and complete all scheduled visits.
7. Subjects who voluntarily decided the participation of the investigation and signed the informed consent.

Exclusion Criteria:

1. Known hypersensitivity or previous allergic reaction to any component of the study devices
2. Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
3. History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
4. History of connective tissue disease.
5. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
6. Subjects who participated in other clinical investigation within 30 days, or in an exclusion period from a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
WSRS grading | 24 weeks after last treatment
  Proportion of responders, defined by at least 1-point improvement from baseline 5-point WSRS, as measured by the blinded live evaluator at 24 weeks after the last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided